CLINICAL TRIAL: NCT05444842
Title: Insulin Iontophoresis Mixed With Oleic Acid Versus Topical Insulin in Patients With Chronic Diabetic Foot Ulcer. Randomized Controlled Trial
Brief Title: Insulin Iontophoresis Mixed With Oleic Acid Versus Topical Insulin in Patients With Chronic Diabetic Foot Ulcer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC/012/003670
Record Dates: First submitted 2022-06-24; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Intervention Model Description: insulin iontophoresis and topical insulin
Who Masked: Participant, Outcomes Assessor
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- insulin iontophoresis (Experimental): the patients will receive insulin iontophoresis for thirty weeks
  Interventions: Other: insulin iontophoresis
- topical insulin (Experimental): the patients will receive topical insulin for thirty weeks
  Interventions: Other: topical insulin
- conventional treatment (Active Comparator): the patients will receive standard dressing and normal saline twice daily for thirty weeks
  Interventions: Other: conventional treatment

INTERVENTIONS:
Other: insulin iontophoresis — All wounds will be thoroughly cleansed with physiologic serum before the therapeutic treatment began (i.e., saline 0.9 percent). after cleaning the wound the insulin ions and oleic acid will be injected into the electrode of iontophoresis device (Phoresor_ IIAuto, ModelPM850, IOMED) then The device was set to the required dose of 40 mA-min, and the current intensity was gradually increased based on the subject's tolerance (ranging from 1 to 4 mA). The device computed the required time for the selected dose automatically.
  Arms: insulin iontophoresis
Other: topical insulin — All wounds will be thoroughly cleansed with physiologic serum before the therapeutic treatment began (i.e., saline 0.9 percent) after cleaning the wound For each 10cm2 of the wound, patients will get ten units (0.1 mL) of insulin crystal in solution with 1mL saline (0.9 percent). An insulin syringe needle was used to spray the solution twice daily on the wound area.
  Arms: topical insulin
Other: conventional treatment — All wounds will be thoroughly cleansed with physiologic serum before the therapeutic treatment began (i.e., saline 0.9 percent) after cleaning the wound For each 10cm2 of wound 1mL 0.9 percent saline was given.
  Arms: conventional treatment

SUMMARY:
This study will be conducted to investigate the effect of Insulin iontophoresis mixed with oleic acid versus topical insulin in patients with chronic diabetic foot ulcer

DETAILED DESCRIPTION:
Despite insulin treatment and a meticulously controlled diet, approximately 15% of all patients with diabetes will, at some time, have non-healing wounds and this is the leading cause of lower extremity amputation. Wound healing involves cell adhesion, migration, proliferation, differentiation, and apoptosis at cellular and molecular levels. Abnormalities of distinct factors of wound healing contribute to defective wound healing in diabetes ulcers, including decreased growth factor production, angiogenic response, macrophage function, collagen accumulation, epidermal barrier.

Insulin has great effect on ulcers healing and tissue regeneration but there is a catch that insulin is a large polymer that have difficulty crossing skin barrier but with using penetration enhancers like oleic acid combined with iontophoresis helps insulin to get through skin especially that affect locally on wound not systematic. Insulin help in restoring the function and structure of the vasculature and improving angiogenesis, reduces the local wound blood glucose concentration, thus reducing the damage resulting from the accumulation of high levels of glucose metabolic intermediates, insulin is the inhibitor of three major proinflammatory transcription factors: Nuclear factor-κB, activator protein-1 and early growth response-1 (EGR-1). insulin relieves the inflammatory response and prevents an excessive inflammatory reaction. Furthermore, insulin inhibits the degradation of immune cell proteins, thus enhancing immune activity. 45 patients with diabetic feet will be assigned randomly into 3 equal group; group A will receive insulin iontophoresis for 13 sessions, group B will receive topical insulin and group C will receive saline dressing for 13 weeks

ELIGIBILITY:
Inclusion Criteria:

* All patients had chronic wound at foot
* The patients ages were ranged from 40 to 70 years
* The subjects were chosen from both sexes
* All patients were diabetic patients

Exclusion Criteria:

* uncontrolled wound bleeding
* severe malnutrition
* severeinfection
* Immunodeficiency
* age>70 years
* renal failure
* liver dysfunction
* ischaemic limbs

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-07-05 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
life disability | up to thirty weeks
  disability of life will be assessed by the quality of life questionnaire; The Questionnaire included 12 main questions, addressing seven specific areas of functional health status (physical functioning, role limitations due to physical health, role limitations due to emotional problems, wound status improvement, social functioning, pain, and general health). All questions were scored on a scale from 0 to 100, with 100 representing the highest level of functioning possible. Aggregate scores were compiled as a percentage of the total points' possible (step 1 chart). The scores from the questions that address a specific area of functional health status were then averaged together, for a final score within each of the dimensions measured (step 2 chart). All seven categories were scored in the same way at the beginning and at the end of the course of care to track the progress of them.
healing rate | up to thirty weeks
  The major goal of this study was to achieve complete wound closure. The main area - final wound area (in mm2/healing time) in days was used to determine the wound healing rate, which was reported as mm2/day